CLINICAL TRIAL: NCT07232537
Title: FINE-REAL Korea: A Non-interventional Study Providing Insights Into the Use of Finerenone in a Routine Clinical Setting in Korea
Brief Title: An Observational Study Called FINE-REAL Korea to Learn More About the Use of the Drug Finerenone in People With Chronic Kidney Disease and Type 2 Diabetes in a Routine Medical Care Setting in South Korea
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23104
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with CKD and T2D: Participants who are newly prescribed finerenone under routine treatment conditions.
  Interventions: Drug: Kerendia (Finerenone, BAY94-8862)

INTERVENTIONS:
Drug: Kerendia (Finerenone, BAY94-8862) — Decision will be taken by the treating physician to initiate treatment with finerenone.

SUMMARY:
This is an observational study in which data from people with chronic kidney disease (CKD) and type 2 diabetes (T2D) who will be receiving finerenone are collected and studied.

Chronic kidney disease is a long-term condition where the kidneys gradually lose their ability to filter waste and extra water from the blood. Type 2 diabetes occurs when the body does not produce enough insulin or does not use it effectively, leading to high blood sugar levels that can harm the kidneys. As a result, CKD can develop as a complication of T2D.

The study drug, finerenone, is already approved for doctors to prescribe to patients with CKD and T2D.

Finerenone is a medication that works by blocking certain proteins known as mineralocorticoid receptors. An increased stimulation of these proteins is thought to damage the kidneys and the heart. By lowering their stimulation, finerenone reduces the risk of kidney disease progressively getting worse.

The main purpose of this study is to learn more about characteristics and treatment patterns of people with CKD and T2D who have recently started or will start finerenone treatment as prescribed by their doctor as part of their routine medical care in South Korea.

The FINE-REAL Korea study is designed to collect additional data on people with CKD and T2D who are treated with finerenone according to the approved product information, and it will work alongside the original FINE-REAL study (NCT05348733) to gather enough information for safety assessments in Korean population.

To achieve this, researchers will collect data on:

* Clinical characteristics of participants, including their medical history related to CKD and T2D, blood pressure, and heart health.
* Reasons for starting finerenone.
* Reasons for stopping finerenone early.
* The planned and actual duration of finerenone treatment.
* The dosing of finerenone.
* Other medications taken alongside finerenone.

The study will also monitor any medical problems (known as adverse events) that participants may experience during the study. All adverse events will be recorded, regardless of whether they are related to the treatment.

One specific concern is hyperkalemia, which refers to high potassium levels in the blood. This condition can occur when finerenone is used with certain blood pressure medications. Researchers want to understand how often hyperkalemia happens and whether it leads to:

* Early discontinuation of finerenone treatment.
* The need for dialysis, a procedure that filters waste from the blood.
* Hospitalization for care.

Data for this study will be collected from medical records and through interviews conducted by study doctors during routine medical visits.

Participants will be involved in the study for up to 12 months, although this duration may be shorter if their finerenone treatment is stopped early.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male participant - All genders (≥18 years old)
* Diagnosis of CKD associated with T2D based on assessment by physician
* Treatment according to local marketing authorization, finerenone 20 or 10 mg. Treatment should have been started up to 8 weeks before or after the ICF is signed.
* Decision to initiate treatment with finerenone must be made before ICF is signed

Exclusion Criteria:

* Participation in an investigational trial at any time during the course of this study
* Contra-indications according to the local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosed of CKD and T2D will be enrolled after the decision for treatment with finerenone has been made by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of clinical characteristics of participants with chronic kidney disease (CKD) and with type 2 diabetes (T2D) | Up to 12 months after start of finerenone
Descriptive summary of reasons for introducing finerenone | Up to 12 months after start of finerenone
Descriptive summary of reasons for discontinuation of finerenone | Up to 12 months after start of finerenone
Planned and actual duration of treatment with finerenone | Up to 12 months after start of finerenone
Planned and actual dosing of finerenone | Up to 12 months after start of finerenone
Descriptive summary of secondary therapies used in participants with CKD and T2D | Up to 12 months after start of finerenone

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) | Up to 30 days after the final treatment with finerenone
  Including treatment emergent adverse events (TEAEs), adverse drug reactions (ADRs), unexpected AEs, unexpected ADRs, serious adverse events (SAEs), and serious adverse drug reactions (SADRs)
Occurrence of hyperkalemia | Up to 30 days after the final treatment with finerenone
  Reported hyperkalemia leading to permanent study drug discontinuation, dialysis or hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access. As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.